CLINICAL TRIAL: NCT06444997
Title: Efficacy and Safety of Oxycodone Hydrochloride and Remifentanil for Long-term Analgesia During Invasive Mechanical Ventilation in Postoperative Patients: A Pilot Study
Brief Title: Efficacy and Safety of Oxycodone Hydrochloride for Long-term Analgesia in ICU Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B2024-161R
Record Dates: First submitted 2024-05-24; First posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Oxycodone; Analgesia; Mechanical Ventilation; Postoperative; Remifentanil
Keywords: Oxycodone; oxycodone hydrochloride; long term analgesic; Analgesia; Mechanical Ventilation; Remifentanil; Pilot Study; ICU
MeSH Terms: conditions — Agnosia | interventions — Oxycodone; Remifentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxycodone Hydrochloride (Experimental): Continuous infusion therapy
  Interventions: Drug: Oxycodone Hydrochloride
- Remifentanil (Active Comparator): Continuous infusion therapy
  Interventions: Drug: Remifentanil

INTERVENTIONS:
Drug: Oxycodone Hydrochloride — Oxycodone hydrochloride will be administered at a continuous infusion dose of 0.03-0.2 mg/kg/h.
  Arms: Oxycodone Hydrochloride
Drug: Remifentanil — Remifentanil will be administered at a continuous infusion dose of 2-9 μg/kg/h.
  Arms: Remifentanil

SUMMARY:
The goal of this clinical trial is to learn if oxycodone hydrochloride works to manage pain in patients requiring mechanical ventilation. It will also assess the safety of oxycodone hydrochloride. The main questions it aims to answer are:

1. Does oxycodone hydrochloride effectively lower the CPOT (Critical Care Pain Observation Tool) score in mechanically ventilated patients?
2. What medical problems do participants have when using oxycodone hydrochloride? Researchers will compare oxycodone hydrochloride to remifentanil to see if oxycodone works better to manage pain in these patients.

Participants will:

* Receive either oxycodone hydrochloride injection at a dose of 0.03-0.2 mg/kg/h or remifentanil injection at a dose of 2-9 μg/kg/h.
* Have their pain scores assessed every 15 minutes until the CPOT score is less than 3. After reaching the target pain score, assessments will be done every 4 hours.
* Have their vital signs and monitoring data recorded.
* Have analgesia and sedation scores recorded from days 1 to 7 after administration, with drug dosages adjusted based on pain scores.
* Have the incidence of adverse reactions and changes in gastrointestinal function observed and recorded from days 1 to 7 after administration.
* If extubated within 7 days, relevant data will be collected based on the time of extubation.
* Be followed up on day 28 through the electronic medical record system to gather data on the extubation success rate and incidence of complications within the 28-day period.

DETAILED DESCRIPTION:
This study is a single-center, single-blind, randomized controlled exploratory study involving subjects aged 18 to 80 who are expected to require mechanical ventilation for ≥24 hours and who were intubated and received mechanical ventilation for less than 3 days before enrollment. Subjects will be treated with either oxycodone hydrochloride injection or remifentanil injection and will be randomly assigned in a 1:1 ratio, giving each subject a 50% chance of being assigned to the control group.

Trial Group: Subjects will receive oxycodone hydrochloride injection at a dose of 0.03-0.2 mg/kg/h. Pain scores will be assessed every 15 minutes until the CPOT (Critical Care Pain Observation Tool) score is less than 3. After achieving the target pain score, pain scores will be assessed every 4 hours.

Control Group: Subjects will receive remifentanil hydrochloride injection at a dose of 2-9 μg/kg/h. Pain scores will be assessed every 15 minutes until the CPOT score is less than 3. After achieving the target pain score, pain scores will be assessed every 4 hours.

During this period, the vital signs and monitoring data of the subjects will be recorded. Analgesia and sedation scores will be recorded from days 1 to 7 after administration, and the analgesic and sedative drug dosages will be adjusted based on the subjects' pain scores. Additionally, the incidence of adverse reactions and changes in gastrointestinal function will be observed and recorded from days 1 to 7 after administration.

There are no biological detection indicators in this study; all evaluations are made by the researchers through scoring sheets and will not affect the subjects' normal treatment. If a subject is extubated and weaned off the ventilator within 7 days, relevant data will be collected based on the time of extubation. On the 28th day after administration, doctors will follow up via the electronic medical record system to gather data on the extubation success rate, incidence of complications, and other relevant indicators within the 28-day period.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤ Age ≤ 80
* Intubated and mechanically ventilated < 3 days prior to enrollment
* Expected need for continuous mechanical ventilation ≥ 24 hours

Exclusion Criteria:

* Patients requiring deep sedation (e.g., mechanical ventilation patients with severe man-machine dyssynchrony, respiratory distress due to severe respiratory failure, application of neuromuscular blockers, status epilepticus, surgical procedures requiring strict immobilization, mild hypothermia treatment, etc.);
* Chronic kidney disease, severe liver dysfunction (Child-Pugh Class C)
* Severe shock requiring norepinephrine ≥ 0.5 µg/kg/min
* American Society of Anesthesiologists (ASA) Class 5 patients (near death)
* Nerve injury or organic pathological changes in the brain
* Need for designated sedatives or anesthetics other than study drug during treatment
* Patients with chronic pain, frequently taking strong opioids, such as morphine
* History of alcohol or drug abuse
* Participation in other opioid studies within 30 days
* Pregnant or lactating women
* Patients with study drug allergy and contraindications Patients who are not suitable for inclusion in the study as judged by the investigator

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of time with Critical care Pain Observation Tool (CPOT) < 3 without rescue analgesia within 7 days of mechanical ventilation. | Mechanical ventilation within 7 days after administration of analgesics.
  By CPOT Form.

SECONDARY OUTCOMES:
Days without mechanical ventilation | Within 28 days after administration
  Collect relevant data by case form
Successful extubation rate | Within 28 days after administration
  Defined as not using non-invasive or invasive mechanical ventilation within 48 hours after the first spontaneous breathing trial (SBT) in 28 days
Ventilator-associated pneumonia | Within 28 days after administration
  Assessed according to diagnostic criteria
Delirium | Within 28 days after administration
  Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). The CAM-ICU provides a binary outcome: the presence or absence of delirium. The assessment results in either a positive or negative diagnosis for delirium, where a positive result indicates the presence of delirium and a worse outcome for the patient.
Length of Stay (LOS) in ICU | From ICU admission to ICU discharge (typically within 1 to 4 weeks)
  Collect relevant data by case form
Change in gastrointestinal function within 7 days of dosing | Postdose 1, 2, 3, 4, 5, 6, 7 days
  Gastrointestinal Failure (GIF) score. The score ranges from 0 to 4, a higher GIF score signifies a more severe gastrointestinal dysfunction and a worse outcome for the patient.
Adverse Event (AE) incidence rate | 7 days postdose
  Investigator assessment by observation

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhong, Principal Investigator — Fudan University
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No